CLINICAL TRIAL: NCT01969565
Title: An Open-label, Single-arm, Phase 1b/ 2 Study of Carfilzomib in Combination With Dexamethasone in Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Study of Carfilzomib in Combination w/Dexamethasone in Patients w/Newly Diagnosed Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Logistical reasons
Sponsor: Emory University (Other)
Collaborators: Onyx Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Jonathan Kaufman, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00060113; ISTCAR511 (Other: Emory University)
Record Dates: First submitted 2013-09-04; First posted 2013-10-25 (Estimated); Results first posted 2015-11-04 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carfilzomib in combination with dexamethasone (Experimental): Carfilzomib will be administered at a dose of 20 mg/m², with a dose escalation to 36 mg/m² after Days 1 and 2 of Cycle 1 in level 1; and at a dose of 20 mg/m², with a dose escalation to 45 mg/m² after Days 1 and 2 of Cycle 1 in level 2 in subjects with multiple myeloma who are newly diagnosed and treatment naïve. Dexamethasone will be given as a fixed dose of 20 mg PO/IV (1, 2, 8, 9, 15, 16, 22, and 23) for cycles 1 to 4 and for subsequent cycles.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib
  Other Names: Kyprolis
Drug: Dexamethasone
  Other Names: Decadron

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of increasing doses of carfilzomib in combination with dexamethasone

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have newly diagnosed multiple myeloma immunoglobulin G (IgG), immunoglobulin A (IgA), immunoglobulin E (IgE) or immunoglobulin D (IgD) by the International Myeloma Foundation (IMF) 2003 Diagnostic Criteria
* Subjects must be treatment naïve.
* Patient must not have been previously treated with any prior systemic therapy for the treatment of multiple myeloma.
* Prior treatment of hypercalcemia or spinal cord compression with corticosteroids does not disqualify the patient (the dose should not exceed the equivalent of 160 mg of dexamethasone in a 2 week period).
* Patients treated with local radiotherapy with or without concomitant exposure to steroids, for pain control or management of cord/nerve root compression, are eligible.
* One week must have lapsed since last date of radiotherapy, which is recommended to be a limited field.
* Patients who require concurrent radiotherapy should have entry to the protocol deferred until the radiotherapy is completed and one week have passed since the last date of therapy.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* All necessary baseline studies for determining eligibility must be obtained within 21 days prior to enrollment.
* Age 18 years at the time of signing Informed Consent.
* Life expectancy of more than three months.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2 or Karnofsky performance status of ≥ 60.
* Subject must be able to adhere to the study visit schedule and other protocol requirements.
* Written informed consent in accordance with federal, local, and institutional guidelines.
* Female subjects of child-bearing potential must have a negative serum pregnancy test within seven days of the first dose and agree to use dual methods of contraception during and for 3 months following last dose of drug.
* Post menopausal females (> 45 years old and without menses for > 1 year) and surgically sterilized females are exempt from a pregnancy test.
* Male subjects must use an effective barrier method of contraception during study and for three months following the last dose if sexually active with a female of child-bearing potential.
* Subjects must be able to receive outpatient treatment and laboratory monitoring at the institute that administers agent.

Exclusion Criteria:

* Patient has > Grade 2 peripheral neuropathy on clinical examination within 14 days before enrollment.
* Renal insufficiency as measured by calculated creatinine clearance < 15 mL/min by Cockroft-Gault formula.
* Subjects with evidence of mucosal or internal bleeding and/or platelet refractory (i.e., unable to maintain a platelet count 50,000 cells/mm³).
* Subjects with an absolute neutrophil count (ANC) < 1000 cells/mm³. Growth factors may not be used to meet ANC eligibility criteria.
* Total bilirubin > 2.0 mg/dL or bilirubin ≥ 2 x upper limit of normal (ULN).
* Subjects with a hemoglobin < 8.0 g/dL (Transfusion are permitted).
* Alanine aminotransferase (ALT) (SGPT) > 2.5 x ULN.
* Aspartate aminotransferase (AST) ≥ 2.5 x ULN.
* Major surgery within three weeks of starting study drug (Cycle 1 Day 1).
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
* Clinically relevant active infection requiring either oral or intravenous antibiotics or antifungal agents.
* Serious co-morbid medical conditions such as chronic obstructive or chronic restrictive pulmonary disease, and cirrhosis.
* Any condition, including laboratory abnormalities, that in the opinion of the Investigator places the subject at unacceptable risk if he/she were to participate in the study.
* Prior malignancy (within the last 3 years) except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ breast cancer, in situ prostate cancer or if the expected survival from other malignancy is less than 90% at 5 years.
* Uncontrolled diabetes mellitus (Fasting Blood Sugar > 400 despite medical treatment).
* Known history of POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M-protein) and skin changes).
* Known HIV infection.
* Known active hepatitis B or C viral infection.
* Plasma cell leukemia.
* Glucocorticoid therapy (prednisone > 20 mg/day or equivalent) within the last three weeks.
* Any prior treatment for multiple myeloma with standard regimens or investigative regimens.
* Subjects with treatment related myelodysplastic syndrome.
* Subjects in whom the required program of oral and intravenous fluid hydration is contraindicated, e.g., due to pre-existing significant pulmonary, cardiac or renal impairment.
* Subjects with known primary amyloidosis.
* Female subject is pregnant or breast-feeding.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Kaufman, MD, Principal Investigator — Emory University
Locations (1):
- Winship Cancer Institute-Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was open to accrual from August 2013 to September 2014.
Pre-assignment Details: One patient consented but withdrew prior to beginning treatment.
Period: Overall Study
Arm/Group | Carfilzomib in Combination With Dexamethasone
Started | 1
Completed | 0
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Carfilzomib in Combination With Dexamethasone
Number analyzed (Participants) | 1
Age, Continuous [Mean (Full Range); unit: years] | 64
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Tolerability and Safety of Increasing Doses of Carfilzomib in Combination With Dexamethasone.
Description: Adverse events will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA) adverse event dictionary. The results will be tabulated to examine their frequency, organ systems affected, and relationship to study treatment. The results of laboratory assessments will be evaluated similarly.
Time Frame: 24 months
Population: Patient withdrew consent before receiving treatment
Groups:
- Carfilzomib in Combination With Dexamethasone: Carfilzomib will be administered at a dose of 20 mg/m2, with a dose escalation to 36 mg/m2 after Days 1 and 2 of Cycle 1 in level 1; and at a dose of 20 mg/m2, with a dose escalation to 45 mg/m2 after Days 1 and 2 of Cycle 1 in level 2 in subjects with multiple myeloma who are newly diagnosed and treatment naïve. Dexamethasone will be given as a fixed dose of 20 mg PO/IV (1, 2, 8, 9, 15, 16, 22, and 23) for cycles 1 to 4 and for subsequent cycles.
  Carfilzomib
  Dexamethasone
Arm/Group | Carfilzomib in Combination With Dexamethasone
Number analyzed (Participants) | 0

2. Primary Outcome: Patients With ≥ VGPR (Very Good Partial Response)
Description: VGPR will be estimated based on the crude proportion of subjects whose best response is Stringent Complete Response (sCR), Complete Response (CR), and VGPR.
Time Frame: 4 months-8 months
Population: Patient withdrew consent before receiving treatment
Arm/Group | Carfilzomib in Combination With Dexamethasone
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Response Rate (ORR), Defined as sCR, CR, Very Good Partial Response (VGPR), and PR at 4 Cycles
Description: The ORR will be estimated based on the crude proportion of subjects for whom best overall response is sCR, CR, VGPR, and PR.
Time Frame: 4 months
Population: Patient withdrew consent before receiving treatment
Arm/Group | Carfilzomib in Combination With Dexamethasone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Carfilzomib in Combination With Dexamethasone
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
One patient consented but withdrew prior to beginning treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes